CLINICAL TRIAL: NCT03149601
Title: Composition and Collection Feasibility of Gut Microbiota in Children With and Without Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Illinois College of Medicine at Peoria (Other)
Responsible Party: Sponsor
Other Study IDs: 1001223
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool samples will be processed and retained for DNA and RNA genomic analysis of microbiome
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Weight: Participants with BMI < 95th percentile
- Obese: Participants with BMI > or = 95th percentile

SUMMARY:
Adults with obesity have an imbalance of bacteria in their intestines which may contribute to weight gain and diseases related to obesity. Restoring the balance of these bacteria (the "microbiota") could help reduce weight and related diseases. However, little is known about this imbalance in children with obesity. This research study will map out the compositions of the gut microbiota of children and compare them with those of children who have healthy weights and different degrees of obesity. This project will also measure the amounts of fatty acids in the stools which are an indication of how efficiently the intestines absorb calories from food. If an imbalance is detected in children with obesity, then this information can help researchers test ways to restore the gut microbiota with hopes of reducing weight and some of its related health problems.

ELIGIBILITY:
Inclusion Criteria:

1) patients aged 5-12 years

Exclusion Criteria:

1. patient who have received either oral or parenteral antibiotics in the last 3 months
2. patients who have a diagnosed immunodeficiency
3. patients who are on medications that modulate the immune system including systemic prednisone and biologics
4. patients who have a gastrointestinal condition which is known to alter the gut flora such as inflammatory bowel disease, chronic diarrhea, celiac disease and eosinophilic gastroenteritis diseases
5. patients who have taken proton pump inhibitors in the last 3 months
6. patients who have taken probiotics in the last 6 months.

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: 150 participants will be recruited from 4 primary care sites (2 urban and two rural) and a tertiary pediatric weight management clinic (PWMC) located in Central Illinois over an 18 month period. Enrollment will equally represent urban and rural lean participant living environments.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota Composition | Over 2 years
  High-throughput sequencing targeting the 16S rRNA gene will be used to detect and identify bacteria in fecal samples. DNA extraction and library preparation will be performed at the University of Illinois College of Medicine at Peoria, and libraries will be subjected to 16S rDNA sequencing (approximately 10k reads will be obtained per sample) on a MiSeq instrument. Using 10k reads per sample provides stable patterns for human stool microbiota. The 16S data will provide information about the presence and abundance of bacteria, and will be analyzed with Qiime, an open source bioinformatics package.
Short Chain Fatty Acid Content | Over 2 years
  Gas Chromatography will be used to measure SCFA amounts, specifically acetate, butyrate, proprionate. Preserved aliquot samples will be analyzed on Agilent GC/MS system (6890GC/5973 MS with 7683B autosampler) with gas chromatography performed on a ZB-WAX (30 m×0.32 mm I.D., 0.25um film thickness) capillary column (Phenomenex, Torrance, CA). The inlet and MSD interface temperatures will both be 250°C, with the ion source temperature adjusted to 230°C. The helium carrier gas will be kept at a constant flow rate of 3.2 ml/min. The temperature program is: initial 2-min isothermal heating at 80°C, followed by an oven temperature increase of 20°C/min to 110°C, then 10°C/min to 130°C, and then 35°C/min to 255°C. Mass spectra will again be recorded in the m/z 50-300 scanning range.
Specimen Quality | Over 2 years
  Technical factors, which may affect microbial compositions (such as times of specimen collection, home freezer storage removal, shipping, and arrival) will be recorded as independent variables. To estimate and minimize the effect of technical variables, principal component analysis will be used and the study will follow the International Human Microbiome Standards

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois College of Medicine at Peoria, Peoria, Illinois, United States